CLINICAL TRIAL: NCT05214443
Title: Per-oral Endoscopic Myotomy With Fundoplication (POEM+F) for Achalasia - a Pilot Study
Brief Title: POEM + F for Achalasia - a Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Hon Chi Yip, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE 2021.648
Record Dates: First submitted 2022-01-15; First posted 2022-01-28 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Achalasia
MeSH Terms: conditions — Esophageal Achalasia | interventions — nephronectin

STUDY DESIGN:
Intervention Model Description: Per-oral endoscopic Myotomy with fundoplication (POEM + F)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- POEM + F arm (Experimental): This arm will receive the POEM + F procedure
  Interventions: Procedure: POEM + F

INTERVENTIONS:
Procedure: POEM + F — POEM would first be performed as per usual technique. Upon completion of the myotomy, a 2cm incision would be created over the adventitial layer at the level of gastro-esophageal junction (GEJ), allowing scope entry into the peritoneal cavity. The anterior part of the gastric fundus would be located, grasped with endoscopic forceps and pulled towards the esophageal myotomy site. The intended anterior fundus would then be anchored to the edge of the muscle at the GEJ, with the use of X-TackTM system. After confirming adequate hemostasis and secure anchorage of fundus to the esophagus, the mucosal entry site for the submucosal tunnel would be closed with endoscopic clips as per usual POEM technique.

SUMMARY:
This is a pilot study to investigate the feasibility of performing per-oral endoscopic Myotomy (POEM) with endoscopic fundoplication for patient with achalasia. Post-POEM reflux is a well documented adverse event after POEM for achalasia. Case series have been published by addition of endoscopic fundoplication procedure during POEM. In the current study, 10 patients would be recruited for investigating the novel POEM procedure with fundoplication by using a new X-tack anchoring device.

DETAILED DESCRIPTION:
Since the first published case series, per-oral endoscopic myotomy (POEM) has emerged as one of the standard treatment options for achalasia. The procedure offers a scarless endoscopic alternative to conventional surgical myotomy. In a recent randomized controlled trial, POEM was found to achieve similar treatment success rate when compared with surgical myotomy. POEM was also found to have reduced serious adverse events. When compared with endoscopic pneumatic dilatation, POEM was demonstrated to have a significantly higher clinical success rate.

One of the major limitations of POEM was the higher incidence of post-procedural acid reflux. During surgical myotomy, a partial fundoplication would routinely be performed to reinforce the gastro-esophageal junction, and such procedure has been proven to reduce post-operative reflux. Multiple studies have confirmed the higher incidence of endoscopic reflux esophagitis and proton pump requirements after POEM than surgical myotomy, including the aforementioned randomized trial.

Modification and standardization of the POEM techniques were proposed to reduce the incidence of reflux esophagitis. Limitation of gastric myotomy length to below 2cm was found to be a useful maneuver. Identification of the two penetrating vessels at cardia may help to correctly measure the length of gastric myotomy, together with the use of double scope technique.

In an attempt to reduce the risk of post-POEM reflux, researchers have also pioneered procedures to mimic surgical fundoplication. The POEM + fundoplication (POEM+F) procedure, was first reported in 2019. It involved anterior myotomy, followed by an anterior partial fundoplication using endoscopic clips and detachable loop. The same group subsequently modified the technique by using a novel endoscopic needle holder device. A recent single-center study reporting results of 25 POEM+F procedures in India also confirmed its reproducibility and safety, as well as a reasonably low incidence of reflux.

A recently developed endoscopic tacking device, X-TackTM (Apollo EndoSurgery, Inc, United States), allows approximation of tissue with the use of a helix tacking system connected to a suture. It could be applied for closure of defect after endoscopic resection. The novel device may also potentially be used for the endoscopic fundoplication by approximating the anterior fundus to the edge of esophageal myotomy during POEM+F. The simple design of the device could make the fundoplication easier and less time consuming. The investigators designed this pilot study to confirm the feasibility of using X-TackTM for POEM+F in patients with achalasia.

ELIGIBILITY:
* Inclusion criteria

  1. Patients with achalasia diagnosed with high resolution manometry, scheduled for elective per-oral endoscopic myotomy
  2. Age >18
* Exclusion criteria

  1. Prior treatment for achalasia, including surgical myotomy, dilatation or POEM.
  2. Prior upper abdominal surgery
  3. Other cases deemed by the examining physician as unsuitable for safe treatment
  4. Patients who refused to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Technical success | 1 day
  Percentage of successful myotomy plus anchorage of gastric fundus to the esophagus by X-TackTM system, without major intra-operative complication.

SECONDARY OUTCOMES:
Clinical success | 1 year
  defined as Eckardt score ≤3
Incidence of symptomatic reflux | 1 year
  Incidence (percentage) of patients with postoperative symptomatic reflux
Incidence of endoscopic esophagitis | 1 year
  Incidence (Percentage) of endoscopic esophagitis, graded according to Los Angeles classification
Adverse events of procedure | 30 days
  Incidence (Percentage) of adverse events related to POEM + F

CONTACTS AND LOCATIONS:
Overall Officials: Hon Chi Yip, FRCSEd, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No